CLINICAL TRIAL: NCT02210663
Title: A Phase 1 Study of Single Agent Veliparib in Japanese Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-489
Record Dates: First submitted 2014-07-25; First posted 2014-08-07 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2016-07

CONDITIONS: Advanced Solid Tumors
Keywords: Breast cancer; PARP; Primary peritoneal cancer; Fallopian tube; Ovarian cancer; veliparib; ABT-888; BRCA
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- veliparib (ABT-888) (Experimental)
  Interventions: Drug: veliparib (ABT-888)

INTERVENTIONS:
Drug: veliparib (ABT-888) — Subjects will be given veliparib twice daily on Days 1-28 every 28 days orally.
  Other Names: veliparib; ABT-888

SUMMARY:
This is a Phase 1 study to evaluate the tolerability, safety, pharmacokinetics and preliminary efficacy of single agent Veliparib in Japanese subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant solid tumor, and any of the following: * Subjects with recurrent high grade serous ovarian cancer who completed or discontinued platinum based therapy; * Subjects with BRCA-mutated breast cancer who have received prior chemotherapy with anthracycline and/or taxanes; * Subjects with deleterious mutations of BRCA with advanced solid tumors who have received available standard therapies.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Life expectancy of greater than 12 weeks.
* Adequate organ and marrow function· Measurable or non-measurable disease.

Exclusion Criteria:

* Major surgery and/or radiation within (<) 4 weeks prior to study enrollment.
* Chemotherapy or hormone therapy within (<) 4 weeks prior to study enrollment except for mitomycin C and nitrosoureas, in which case it is 6 weeks.
* Any investigational agents within (<) 4 weeks prior to study enrollment.
* Any anti-cancer Chinese medicine/herbal remedies within 14 days prior to study enrollment.
* Toxicities (with the exception of alopecia) from prior major surgery, radiation, or systemic chemotherapy have not recovered to less than grade 2.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities of veliparib | During the first cycle (28 days) of veliparib administration

SECONDARY OUTCOMES:
Change in participant physical exam measurements | Approximately 1 year
  Blood pressure, pulse and body temperature
Change in participant clinical lab results | Approximately 1 year
  Hematology, Chemistry and Urinalysis
Number of participants with adverse events | Approximately 1 year
  Collect all adverse events at each visit and assess according to National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03
Preliminary tumor response | Participants will be followed for the duration of an expected average of 8 months.
  According to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1
Maximum observed plasma concentration (Cmax) | For 24 hours following veliparib dosing.
  Maximum observed concentration, occurring at Tmax
The time to Cmax (peak time, Tmax) | For 24 hours following veliparib dosing.
  The time at which maximum plasma concentration (Cmax) is observed.
The area under the plasma concentration-time curve (AUC) | For 24 hours following veliparib dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Hideyuki Hashiba, BS, Study Director — AbbVie
Locations (3):
- Japan (3):
  - Site Reference ID/Investigator# 128056, Hidaka-shi
  - Site Reference ID/Investigator# 129976, Hyōgo
  - Site Reference ID/Investigator# 128057, Tokyo

REFERENCES:
- [Result] Nishikawa T, Matsumoto K, Tamura K, Yoshida H, Imai Y, Miyasaka A, Onoe T, Yamaguchi S, Shimizu C, Yonemori K, Shimoi T, Yunokawa M, Xiong H, Nuthalapati S, Hashiba H, Kiriyama T, Leahy T, Komarnitsky P, Fujiwara K. Phase 1 dose-escalation study of single-agent veliparib in Japanese patients with advanced solid tumors. Cancer Sci. 2017 Sep;108(9):1834-1842. doi: 10.1111/cas.13307. Epub 2017 Aug 5. PMID 28665051